CLINICAL TRIAL: NCT04103515
Title: In Vivo Determination of Knee Kinematics for Subjects Having a Zimmer-Biomet Persona PCR or PS TKA
Brief Title: Knee Kinematics for Subjects With Zimmer-Biomet Posterior Cruciate Retaining or Posterior Stabilizing Total Knee Arthroplasty
Acronym: PCR PS TKA
Status: Completed | Type: Observational
Sponsor: The University of Tennessee, Knoxville (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Principal Investigator, Richard Komistek, Principal Investigator, The University of Tennessee, Knoxville
Other Study IDs: WIRB20183083
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Results first posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Arthroplasty, Replacement, Knee; Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Subjects implanted with PCR TKA: Subjects who have been implanted with a Zimmer-Biomet Posterior Cruciate Retaining total knee arthroplasty
  Interventions: Device: Zimmer-Biomet Posterior Cruciate Retaining total knee arthroplasty
- Subjects implanted with PS TKA: Subjects who have been implanted with a Zimmer-Biomet Posterior Stabilizing total knee arthroplasty
  Interventions: Device: Zimmer-Biomet Posterior Stabilizing total knee arthroplasty

INTERVENTIONS:
Device: Zimmer-Biomet Posterior Cruciate Retaining total knee arthroplasty — Zimmer-Biomet Posterior Cruciate Retaining total knee arthroplasty
  Groups: Subjects implanted with PCR TKA
Device: Zimmer-Biomet Posterior Stabilizing total knee arthroplasty — Zimmer-Biomet Posterior Stabilizing total knee arthroplasty
  Groups: Subjects implanted with PS TKA

SUMMARY:
25 subjects implanted with a Zimmer-Biomet Posterior Cruciate Retaining (PCR) total knee arthroplasty (TKA) and 25 subjects implanted with a Zimmer-Biomet Posterior Stabilizing (PS) TKA will be asked to perform stepping up and deep knee bend activities while under fluoroscopic surveillance (x-ray video). The movements between the two different types of TKAs will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will have a Zimmer Persona PCR or PS TKA.
* Subjects must be at least six months post-operative.
* Subjects will have KSS greater than 75.
* Participants must be able to perform the required activities - stepping up and a deep knee bend.
* Subjects must be willing to sign the Informed Consent (IC) / HIPAA form to participate in the study.
* Bilateral subjects may be included in the subject population

Exclusion Criteria:

* Pregnant, potentially pregnant or lactating females. To satisfy radiation protocol, each female subject will be asked if she is pregnant, or possibly could be pregnant. A pregnant person will not be allowed to participate in the study. To ensure this, a pregnancy test will be administered to any female participants of child bearing age who have not had a hysterectomy.
* Subjects without the required type of knee implant.
* Subjects who are unable to perform stepping up and deep knee bend.
* Subjects who are unwilling to sign Informed Consent/HIPAA documents.
* Subjects who do not speak English and/or French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients implanted with a Zimmer-Biomet posterior cruciate retaining (PCR) or Zimmer-Biomet posterior stabilizing total knee arthroplasty (TKA)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2020-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Komistek, PhD, Principal Investigator — University of Tennessee
Locations (3):
- United States (2):
  - Rothman Institute, Bryn Mawr, Pennsylvania
  - University of Tennessee, Knoxville, Tennessee
- The Institute for Locomotion, Aix-Marseille University, Hopital Sainte-Marguerite, Marseille, France

IPD SHARING:
Plan to Share IPD: No
Researchers would like to retain this study data in our secure database so as to continue to add relevant, current data to our digital collection to help us work with manufacturers in the future to create better implants that last longer and will not require revision surgery. Participants will be asked if their study data may remain a part of the University of Tennessee's Center for Musculoskeletal Research data collection for use in future studies in the IC. Identifiers are automatically removed from the database upon entry into the secure server. Data shared with sponsors is de-identified.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Subjects Implanted With PCR TKA | Subjects Implanted With PS TKA
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Subjects Implanted With PCR TKA | Subjects Implanted With PS TKA | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 16 | 29
  Male | 12 | 9 | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Lateral Condyle Kinematic Translations - Step up
Description: Lateral Condyle Kinematics Translations during stepping up activity. Data represents the motion of a specific part of the femur bone (in this case lateral femoral condyle) during the specified activity (in this case a step up). The kinematics (motion) is measured from the beginning of the activity to the end of the activity. Positive represents anterior motion of the femur, and negative represents posterior rollback of the femur. Data is only collected at a single time point and therefore refers to the motion of the femur bone during a specific activity at a single point in time.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Subjects Implanted With PCR TKA | Subjects Implanted With PS TKA
Number analyzed (Participants) | 25 | 25
mm | 1.15 (3.03) | 2.28 (3.42)

2. Primary Outcome: Lateral Condyle Kinematics Translations - Deep Knee Bend
Description: Lateral Condyle Kinematics Translations during deep knee bend activity. Data represents the motion of a specific part of the femur bone (in this case lateral femoral condyle) during the specified activity (in this case a deep knee bend). The kinematics (motion) is measured from the beginning of the activity to the end of the activity. Positive represents anterior motion of the femur, and negative represents posterior rollback of the femur. Data is only collected at a single time point and therefore refers to the motion of the femur bone during a specific activity at a single point in time.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Subjects Implanted With PCR TKA | Subjects Implanted With PS TKA
Number analyzed (Participants) | 25 | 25
mm | -1.52 (2.09) | -6.80 (3.47)

3. Primary Outcome: Medial Condyle Kinematics Translations - Step Up
Description: Medial Condyle Kinematics Translations during stepping up activity. Data represents the motion of a specific part of the femur bone (in this case medial femoral condyle) during the specified activity (in this case a step up). The kinematics (motion) is measured from the beginning of the activity to the end of the activity. Positive represents anterior motion of the femur, and negative represents posterior rollback of the femur. Data is only collected at a single time point and therefore refers to the motion of the femur bone during a specific activity at a single point in time.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Subjects Implanted With PCR TKA | Subjects Implanted With PS TKA
Number analyzed (Participants) | 25 | 25
mm | -0.36 (2.97) | 0.16 (3.91)

4. Primary Outcome: Medial Condyle Kinematics Translations - Deep Knee Bend
Description: Medial Condyle Kinematics Translations during deep knee bend activity. Medial Condyle Kinematics Translations during stepping up activity. Data represents the motion of a specific part of the femur bone (in this case medial femoral condyle) during the specified activity (in this case a deep knee bend). The kinematics (motion) is measured from the beginning of the activity to the end of the activity. Positive represents anterior motion of the femur, and negative represents posterior rollback of the femur. Data is only collected at a single time point and therefore refers to the motion of the femur bone during a specific activity at a single point in time.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Subjects Implanted With PCR TKA | Subjects Implanted With PS TKA
Number analyzed (Participants) | 25 | 25
mm | 0.13 (2.09) | -4.25 (3.32)

ADVERSE EVENTS:
Time Frame: Baseline. Data is collected only on a single day, and no participant follow-up was collected. Thus, this section describes whether or not there were any adverse events on the single day of data collection
Arm/Group | Subjects Implanted With PCR TKA | Subjects Implanted With PS TKA
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-01-03): https://cdn.clinicaltrials.gov/large-docs/15/NCT04103515/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-03): https://cdn.clinicaltrials.gov/large-docs/15/NCT04103515/SAP_001.pdf